CLINICAL TRIAL: NCT03838367
Title: A Phase Ib/II Study of Leronlimab (PRO 140) Combined With Carboplatin in Patients With CCR5+ Metastatic Triple Negative Breast Cancer (mTNBC)
Brief Title: Leronlimab (PRO 140) Combined With Carboplatin in Patients With Cytokine Chemokine Receptor 5 Positive (CCR5+) mTNBC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated prematurely due to business reasons. Participants are no longer examined or receiving intervention.
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD07_TNBC
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: TNBC; PRO 140
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — leronlimab; Carboplatin; Maximum Tolerated Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I-Cohort A: 350 mg PRO 140 SC weekly + AUC 5 Carboplatin (Experimental): Cohort A: 350 mg PRO 140 SC weekly + AUC 5 Carboplatin every 3 weeks
  Interventions: Drug: 350 mg leronlimab; Drug: AUC 5 Carboplatin
- Phase I-Cohort B: 525 mg PRO 140 SC weekly + AUC 5 Carboplatin (Experimental): Cohort B: 525 mg PRO 140 SC weekly + AUC 5 Carboplatin every 3 weeks
  Interventions: Drug: 525 mg leronlimab; Drug: AUC 5 Carboplatin
- Phase I-Cohort C: 700 mg PRO 140 SC weekly + AUC 5 Carboplatin (Experimental): Cohort C: 700 mg PRO 140 SC weekly + AUC 5 Carboplatin every 3 weeks
  Interventions: Drug: 700 mg leronlimab; Drug: AUC 5 Carboplatin
- Phase II- MTD to be established for the combination treatment (Experimental): MTD PRO 140 SC + AUC 5 Carboplatin
  Interventions: Drug: AUC 5 Carboplatin; Drug: Maximum Tolerated Dose (MTD) of leronlimab

INTERVENTIONS:
Drug: 350 mg leronlimab — leronlimab is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: PRO 140
  Arms: Phase I-Cohort A: 350 mg PRO 140 SC weekly + AUC 5 Carboplatin
Drug: 525 mg leronlimab — leronlimab is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: PRO 140
  Arms: Phase I-Cohort B: 525 mg PRO 140 SC weekly + AUC 5 Carboplatin
Drug: 700 mg leronlimab — leronlimab is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: PRO 140
  Arms: Phase I-Cohort C: 700 mg PRO 140 SC weekly + AUC 5 Carboplatin
Drug: AUC 5 Carboplatin — Carboplatin is an anticancer drug chemotherapy drug.
  Other Names: Paraplatin
Drug: Maximum Tolerated Dose (MTD) of leronlimab — The decision on the MTD will be made following the results obtained from Phase I studies
  Other Names: PRO 140
  Arms: Phase II- MTD to be established for the combination treatment

SUMMARY:
This is a phase Ib/II Study of Leronlimab (PRO 140) combined with Carboplatin in Patients with CCR5+ Metastatic Triple Negative Breast Cancer (mTNBC).

Study population will consist of patients with CCR5-positive, locally advanced or metastatic triple-negative breast cancer (mTNBC) who are naïve to chemotherapy in metastatic setting but have been exposed to anthracyclines and taxane in neoadjuvant and adjuvant settings (first-line).

DETAILED DESCRIPTION:
Phase Ib

Phase Ib is a dose escalation phase with 3 dose levels (cohorts) of leronlimab (PRO 140) administered in combination with a fixed dose of carboplatin at AUC 5 (area under the curve). This dose finding portion of study will follow a "3+3" designed to determine the maximum tolerated dose (MTD) of leronlimab (PRO 140) administered as subcutaneous (SC) injection in subjects with histologically confirmed mTNBC that express CCR5.

Phase II

Phase II is a single arm study with 30 patients in order to test the hypothesis that the combination of carboplatin AUC 5 intravenously and MTD of leronlimab (PRO 140) SC will increase Progression Free Survival (PFS) in patients with CCR5 + mTNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically confirmed diagnosis of TNBC. Must demonstrate HER-2 negative (IHC 0, 1+, or fluorescence in situ hybridization (FISH) negative and ER<1%, and PR < 1%, per ASCO/CAP criteria);
2. Demonstrate CCR5 + by IHC (>10% membranous staining completed at the reference laboratory of Dr. Hallgeir Rui at Medical College of Wisconsin).

   Note: This test will be done as part of the pre-screening period. It will be performed in archival metastatic tissue. If archival tissue is not available then, fresh biopsy will be done;
3. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (in case archival tissue is not available);
4. Patients with stage IV de-novo disease or patients that develop recurrence after completion of neoadjuvant or adjuvant therapy are eligible; Note: Patients who have been exposed to carboplatin in neoadjuvant or adjuvant setting will be allowed to enroll, if they have progressed ≥ 6 months from completion of treatment.
5. Phase 1 study section:

   Subjects must have disease recurrence and progression after ≤ 2 line of therapy in metastatic setting but untreated with carboplatin;

   Phase 2 study section:

   Subjects must be naive to chemotherapy or untreated with carboplatin in metastatic setting (first-line) OR excluding carboplatin chemotherapy, subjects must have failed first-line combination of chemotherapy and a checkpoint inhibitor in metastatic setting;
6. Patients must have measurable disease based on RECIST v1.1;
7. Female patients, ≥ 18 years of age;
8. Patients must exhibit a/an ECOG performance status of 0-1;
9. Life expectancy of at least 6 months;
10. Patients must have adequate organ and bone marrow function within 28 days prior to registration, as defined below:

    * leukocytes ≥ 3,000/mcL;
    * absolute neutrophil count ≥ 1,500/mcL;
    * platelets ≥ 100,000/mcL;
    * total bilirubin: within normal institutional limits;
    * AST(SGOT) &ALT(SPGT) ≤ 2.5 X institutional upper limit of normal (ULN) (applicable to all patients, irrespective of liver disease or metastasis); and
    * creatinine: within normal institutional limits.
11. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
12. Females of child-bearing potential (FOCBP) and males must agree to use two medically accepted methods of contraception with hormonal or barrier method of birth control, or abstinence, prior to study entry, for the duration of study participation and for 60 days after the last dose of study drug (Refer to Appendix 1). Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Note: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; and
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
13. FOCBP must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
14. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

1. HER-2 overexpressed/amplified metastatic breast cancer (MBC) (Appendix 2 for guidelines from ASCO);
2. ER and or PR expressing tumors;
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days prior to enrollment;
4. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible;
5. Patients who have had prior exposure to CCR5 antagonists are not eligible;
6. Patients who have a known additional malignancy that is progressing or requires active treatment are not eligible. Patients who have had a prior diagnosis of cancer and if it has been <3 years since their last treatment are not eligible. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
7. Has an active infection requiring systemic therapy. Note: Patients must complete any treatment with antibiotics prior to registration;
8. Patients who have a known HIV positive status or known/ active Hepatitis B and/or C infection are not eligible;
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial; and
12. Is pregnant or breastfeeding, or expecting to conceive or have children within the projected duration of the trial, starting with the pre-screening or screening visit through the duration of study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients, >=18 years of age;
Enrollment: 10 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Study Director — CytoDyn, Inc.
Locations (2):
- United States (2):
  - Quest Clinical Research, San Francisco, California
  - CD07 Investigational Site, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was early terminated, and no participants were enrolled to the Phase II arm of the trial.
Period: Overall Study
Arm/Group | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase II- MTD to be Established for the Combination Treatment
Started | 3 | 4 | 3 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 0
Not completed — Early termination of study | 3 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of leronlimab (PRO 140) were included in the baseline analysis population. Study was early terminated and no participants were enrolled to the Phase II arm of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase II- MTD to be Established for the Combination Treatment | Total
Number analyzed (Participants) | 3 | 4 | 3 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 3 | 3 | 2 |  | 8
  >=65 years | 0 | 1 | 1 |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.67 (7.76) | 55.75 (11.32) | 61.67 (8.73) |  | 53.30 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 |  | 10
  Male | 0 | 0 | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 |  | 0
  Not Hispanic or Latino | 2 | 4 | 3 |  | 9
  Unknown or Not Reported | 1 | 0 | 0 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 1 | 1 | 0 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 |  | 0
  White | 1 | 3 | 3 |  | 7
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 0 | 0 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 |  | 10
Height [Mean (Standard Deviation); unit: cm] — Population: No height data was collected for 2 participants.
  cm
    number analyzed (Participants) | 2 | 4 | 2 | 0 | 8
    (all) | 160.05 (2.55) | 162.85 (6.23) | 164.30 (3.30) |  | 162.51 (5.11)
Weight [Mean (Standard Deviation); unit: kg] — Population: No weight data was collected from 1 participant.
  kg
    number analyzed (Participants) | 3 | 4 | 2 | 0 | 9
    (all) | 85.73 (32.08) | 66.50 (3.54) | 82.90 (11.40) |  | 76.60 (21.44)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: No data was collected from 2 participants.
  kg/m2
    number analyzed (Participants) | 2 | 4 | 2 | 0 | 8
    (all) | 24.64 (0.96) | 25.09 (0.91) | 30.58 (3.00) |  | 26.35 (2.98)

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Leronlimab (PRO 140) When Combined With Carboplatin AUC5
Description: The MTD is defined as 1 dose level (cohort) below the dose in which dose limiting toxicities (DLTs) were observed in >= 33% of the participants.
Time Frame: From treatment cycle 1 day 1 (C1D1) until MTD reached (each cycle being 3 weeks), up to 26 weeks
Population: The Intent-to-Treat (ITT) population (N=10) consists of all subjects who received at least one dose of leronlimab (PRO 140) and have measurable disease at baseline. The calculation of the sample size is based on the traditional 3+3 dose escalation scheme.
Measure: Number; unit: mg
Groups:
- Phase 1b: Including 3 Dose Levels (Cohort A, Cohort B, and Cohort C): Phase 1b is a dose escalation phase with 3 dose levels (cohorts) of leronlimab (PRO 140) administered in combination with a fixed dose of carboplatin at AUC 5.
Arm/Group | Phase 1b: Including 3 Dose Levels (Cohort A, Cohort B, and Cohort C)
Number analyzed (Participants) | 10
mg | 700

2. Primary Outcome: Phase II: Progression Free Survival (PFS) Defined as Time in Months From the Date of First Study Treatment to the Date of Disease Progression or Death From Any Cause, Whichever Comes First.
Description: All patients who received at least one dose of leronlimab (PRO 140) and carboplatin combination was intended to be included in the primary analyses of PFS. The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria was planned to be used for objective tumor response assessment.
Time Frame: Planned every 6 to 9 weeks after Phase II study start, until progression or death, assessing up to 2 years after completion of treatment
Population: No subjects were enrolled in the Phase II portion of the trial due to early termination of the study. No data was collected for this outcome measure.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase I: Number of Participants With Any Adverse Events (AE) or Serious Adverse Events (SAE) Collected From the Time of First Treatment Until Study Termination to Evaluate Safety of Leronlimab (PRO 140) and Carboplatin in Subjects With CCR5+ mTNBC.
Description: For Phase I: Adverse events followed National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. This will be the Number of Participants with Any Adverse Events (AE) or Serious Adverse Events (SAE) collected from the time of first treatment until study termination to evaluate safety of leronlimab (PRO 140) and carboplatin in subjects with CCR5+ metastatic triple negative breast cancer.
Time Frame: From Cycle 1, Day 1 (each treatment cycle is 3 weeks) until last dose of study drug, up to 26 weeks
Population: The safety population consists of all subjects who received at least one dose of leronlimab (PRO 140).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin
Number analyzed (Participants) | 3 | 4 | 3
Participants
  Participants with any AEs | 3 | 4 | 2
  Participants with any SAEs | 1 | 1 | 0

4. Secondary Outcome: Phase II: Progression Free Survival (PFS) According to RECIST v1.1 in Participants With Detectable Programmed Death-Ligand 1 (PD-L1)
Description: Phase II: Progression Free Survival (PFS) according to RECIST v1.1 in participants with Detectable Programmed Death-Ligand 1 (PD-L1)
  Trial was terminated prematurely and no efficacy data was collected from the Phase II portion.
Time Frame: as for outcome 2
Population: No subjects were included in this outcome measure due to early termination of the trial.
Groups:
- Phase II- MTD to be Established for the Combination Treatment: The trial was terminated prematurely and no efficacy data is available.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase II: Overall Response Rate (ORR, Defined as Complete Response (CR) + Partial Response (PR)), and Clinical Benefit Rate (CBR, Defined as CR + PR + Stable Disease (SD)) in Subjects With CCR5+ mTNBC Treated With Leronlimab (PRO 140) and Carboplatin.
Description: Phase II: Overall response rate (ORR, defined as Complete Response (CR) + Partial Response (PR)), and clinical benefit rate (CBR, defined as CR + PR + Stable Disease (SD)) in subjects with CCR5+ mTNBC treated with
  The trial was terminated early, efficacy data is not available
Time Frame: as for outcome 2
Population: Study was terminated early, no safety data was collected.
Arm/Group | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Phase II: Time to New Metastases (TTNM)
Description: Trial was terminated prematurely and no efficacy data was collected.
Time Frame: as for outcome 2
Population: No subjects were included in this outcome measure due to early termination of the trial.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase II: The Change From Baseline in Circulating Tumor Cells (CTC) Level in the Peripheral Blood.
Description: Phase II: The change from baseline in circulating tumor cells (CTC) level in the peripheral blood.
  No efficacy data was available due to early termination of the trial.
Time Frame: Planned every 21 days (i.e., Day 1 of each treatment cycle) through treatment completion, an average of 6 months.
Population: No subjects were included in this outcome measure due to early termination of the trial.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase II: Overall Survival Defined as Time in Months From the Date of First Study Treatment to the Date of Death;
Description: Phase II: Overall survival defined as time in months from the date of first study treatment to the date of death; No efficacy data is available due to early termination of the trial.
Time Frame: Planned from Day 1 to death from any cause, assessing up to 2 years after completion of treatment.
Population: No subjects were included in this outcome measure due to early termination of the trial.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase II: Number, Frequency, and Severity of AEs Collected From the Time of First Treatment Until 12 Weeks After Study Treatment Completion to Evaluate Safety of Leronlimab (PRO 140) and Carboplatin in Subjects With CCR5+ mTNBC.
Description: Phase II: Number, frequency, and severity of AEs collected from the time of first treatment until 12 weeks after study treatment completion to evaluate safety of leronlimab (PRO 140) and carboplatin in subjects with CCR5+ mTNBC.
  No safety data was available from the Phase II portion of the trial due to early termination of the study.
Time Frame: Planned from Cycle 1, Day 1 (each treatment cycle is 21 days) to 12 weeks after the last dose of study drug)
Population: No subjects were included in this outcome measure due to early termination of the trial.
Arm/Group | Phase II- MTD to be Established for the Combination Treatment
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Measure Immune Biomarkers (PD-L1) in CTCs, Metastatic Tissue and Immune Cells Such as Cancer Associated Macrophage-like Cells (CAMLs) and Correlate With Therapeutic Benefit (PFS)
Description: Measure immune biomarkers (PD-L1) in CTCs, metastatic tissue and immune cells such as CAMLs and correlate with therapeutic benefit (PFS) No subjects were included in this outcome measure due to early termination of the trial.
Time Frame: Planned every 21 days (i.e., Day 1 of each treatment cycle) through treatment completion, an average of 6 months.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Correlation Between CCR5 Expression (CTCs, CAMLs) and PD- L1 Expression.
Description: No subjects were included in this outcome measure due to early termination of the trial.
Time Frame: Planned every 21 days (i.e., Day 1 of each treatment cycle) through treatment completion, an average of 6 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of first treatment until the early termination of the study to evaluate safety of leronlimab (PRO 140) and carboplatin in subjects with CCR5+ mTNBC (up to approximately 30 months).
Description: Safety were assessed by close monitoring and timely assessment of adverse events, laboratory parameters (blood tests, urinalysis), vital signs Blood pressure, heart rate), subject's medical condition (physical examination including weight), general well-being and activities of daily life (Eastern Cooperative Oncology Group (ECOG) performance status).
Arm/Group | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin | Phase II- MTD to be Established for the Combination Treatment
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=3) | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=4) | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=3) | Phase II- MTD to be Established for the Combination Treatment (N=0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I-Cohort A: 350 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=3) | Phase I-Cohort B: 525 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=4) | Phase I-Cohort C: 700 mg PRO 140 SC Weekly + AUC 5 Carboplatin (N=3) | Phase II- MTD to be Established for the Combination Treatment (N=0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Temporary Reddening of Skin
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (5) | 4 (6) | 1 (1) | 0 (0) — Verbatim term: Fatigue; Fatigue R/T Insomnia; Light Fatigue
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Verbatim term: Sore Throat
Lymph Gland Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Allergic Reaction to Carboplatin Infusion
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Verbatim term: Lightheaded; dizziness
Injection Site Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Bruise at left injection site/ Bruising at right and left injection site
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Indigestion
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Mood Swings (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Metallic Taste in Mouth
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Fever
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Verbatim term: Body aches/ general pain
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Decreased (Investigations) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Verbatim term: BL GI Disorder Other: Diverticulitis
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Verbatim term: Bloating
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Trial was terminated prematurely prior to Phase II section of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03838367/Prot_002.pdf
  • Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03838367/SAP_003.pdf